CLINICAL TRIAL: NCT03620188
Title: Are we Meeting Patient Treatment Goals With Guideline-based Therapy for Psoriatic Arthritis
Brief Title: Treatment Goals in Psoriatic Arthritis
Acronym: PaGoPsA
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: IRB00184580
Record Dates: First submitted 2018-08-03; First posted 2018-08-08 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Psoriatic Arthritis
Keywords: Patient treatment goals
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Standard of care — Standard of care in PsA is outline in treatment guidelines as adjustment of therapy every 3 months until goals of treatment are being met. Goals of treatment are defined as remission or low disease activity.

SUMMARY:
The PaGoPsA study objective is to ascertain if guideline-based psoriatic arthritis clinical care achieves individual patient goals as articulated by patients, and to identify predictors of achieving individual patient goals from psoriatic arthritis treatment.

DETAILED DESCRIPTION:
Psoriatic arthritis (PsA) is a heterogeneous autoimmune disease that occurs in one in three people with the skin disease psoriasis. PsA can cause arthritis (joint inflammation), enthesitis (tendon and ligament inflammation), sausage digits (swollen entire finger or toe), spondyloarthritis (spinal inflammation). Skin involvement by psoriasis is also highly variable in terms of psoriasis type and location. Through combined skin and musculoskeletal involvement, psoriatic disease has a significant life impact with decrease quality of life including uncomfortable symptoms, ability to participate in life and functioning. Medications used to treat PsA have sometimes an uneven effect on the various PsA manifestations where some are more effective for skin while others more effective for the joints. In this context, clinical care and treatment of PsA is a complex process which balances disease activity with medication risks and benefits as well as patient priorities. Professional PsA treatments guidelines state that PsA treatment goals are disease remission or low disease activity. Several studies to date have shown that physicians tend to overestimate remission and low disease activity in PsA patients when compared to disease activity indices. Also patients and physicians frequently do not align on perceptions of remission or low disease activity. In the proposed study the investigators aim to identify predictors of successful treatment from a patient perspective on a range of disease measures including psoriasis, arthritis, enthesitis, dactylitis, patient reported outcomes, and laboratory assessments which are routinely collected in the clinical care of PsA. Secondary endpoints are to quantify longitudinally how stable a state of treatment success is from a patient perspective, and to define score ranges for disease measurements, including health-related quality of life measures, that correspond to treatment success from a patient perspective. The impact of this research is that the investigators will be able to define parameters predictive of achieving treatment success from a patient perspective, which will then inform goals of care for psoriatic arthritis.

ELIGIBILITY:
Inclusion Criteria:

* English speaking/reading adults
* Patients of the Johns Hopkins Arthritis Center and/or the Johns Hopkins Psoriatic Arthritis Clinical Program
* Followed every 3-4 months for regular psoriatic arthritis clinical care
* Meet Classification Criteria for Psoriatic Arthritis (CASPAR)
* Able to interact with touch screen computer.

Exclusion Criteria:

None

Ages: 18 Years to 95 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults with a diagnosis of psoriatic arthritis meeting CASPAR classification criteria for psoriatic arthritis who are followed every 3-4 months for regular rheumatologic care. Consecutive clinic patients will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2018-12-20 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Predictors of reaching PsA treatment goals/treatment success from a patient perspective. | 12-16 weeks
  The primary outcome determination is based on the patients' report of whether they are/are not at goal with their PsA treatment.

SECONDARY OUTCOMES:
To define a status of PsA treatment where patient treatment goals have been met. | 52 weeks
  Score ranges that correspond to a status of patients' treatment goals met on a set of PsA outcome measures used in the study, including composite disease activity measures.
Improvement thresholds (treatment success) that correspond to a patient transition from goals not met to met. | 12-16 weeks
  Meaningful change values in patients who transition longitudinally from goals not met to goals met.
Worsening thresholds (treatment failure) if transition is from goals met to not met. | 12-16 weeks
  Meaningful change values in patients who transition longitudinally from goals met to goals not met disease activity categories.
Prevalence of treatment success in guideline -based treatment in psoriatic arthritis from the patients' perspective | 52 weeks
  Prevalence of patients reporting they met PsA treatment goals (successful treatment) from their perspective.
Stability of a state of treatment goals met at subsequent study visits. | 52 weeks
  Frequency and direction of longitudinal transitions between treatment goals/met not met states: 3 observations/participant.

CONTACTS AND LOCATIONS:
Overall Officials: Ana-Maria Orbai, MD, MHS, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Orbai AM, de Wit M, Mease P, Shea JA, Gossec L, Leung YY, Tillett W, Elmamoun M, Callis Duffin K, Campbell W, Christensen R, Coates L, Dures E, Eder L, FitzGerald O, Gladman D, Goel N, Grieb SD, Hewlett S, Hoejgaard P, Kalyoncu U, Lindsay C, McHugh N, Shea B, Steinkoenig I, Strand V, Ogdie A. International patient and physician consensus on a psoriatic arthritis core outcome set for clinical trials. Ann Rheum Dis. 2017 Apr;76(4):673-680. doi: 10.1136/annrheumdis-2016-210242. Epub 2016 Sep 9. PMID 27613807
- See also: Prior work on patient priorities for psoriatic arthritis treatment — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5344772/

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-09-25): https://cdn.clinicaltrials.gov/large-docs/88/NCT03620188/Prot_SAP_000.pdf
  • Informed Consent Form (2020-05-12): https://cdn.clinicaltrials.gov/large-docs/88/NCT03620188/ICF_001.pdf